CLINICAL TRIAL: NCT02643823
Title: Safety and Efficacy Study of Human Umbilical Cord-Mesenchymal Stem Cells for Rheumatoid Arthritis
Brief Title: Human Umbilical Cord-Mesenchymal Stem Cells for Rheumatoid Arthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Futian People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-Rheumatoid Arthritis
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Human Umbilical Cord Mesenchymal Stem Cell; Mesenchymal Stem Cell; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents; Anti-Inflammatory Agents, Non-Steroidal; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hUC-MSC + DMARDs (Experimental): Patients will be treated in combination with hUC-MSC and DMARDs with a 12 months follow-up.
  Interventions: Biological: hUC-MSC + DMARDs
- DMARDs (Active Comparator): Patients will be treated by Rheumatoid Arthritis With Disease-Modifying Drugs (DMARDs) with a 12 months follow-up.
  Interventions: Drug: DMARDs

INTERVENTIONS:
Biological: hUC-MSC + DMARDs — Patients will be treated by conventional drugs (DMARDs) for alleviating disease. Combinated with a single dose of 2×107 hUC-MSC will treated to patients, IV, Repeat every weeks for four times.
  Other Names: Human Umbilical Cord-Mesenchymal Stem Cells
  Arms: hUC-MSC + DMARDs
Drug: DMARDs — Patients will be treated by conventional drugs (DMARDs) for alleviating disease.
  Other Names: NSAIDs; Methotrexate
  Arms: DMARDs

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cell(hUC-MSC) for Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Human umbilical cord mesenchymal stem cells exhibit the potential to differentiate into chondrocyte and osteocyte, which have been confirmed in in vivo and in vitro experiments. There have been few clinical reports describing umbilical cord mesenchymal stem cells for treatment of Rheumatoid Arthritis.

To investigate the effects of hUC-MSC treatment for Rheumatoid Arthritis, 20 patients with Rheumatoid Arthritis will be enrolled and receive 4 times of hUC-MSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 Rheumatoid Arthritis patient;
* Patients must consent in writing to participate in the study by signing and dating an informed consent document;
* Patients must have a diagnosis of Rheumatoid Arthritis according to the 2010 ACR/EULAR criteria for at least 12 weeks duration;
* Stage I and II according to X-ray.

Exclusion Criteria:

* History of neurological disease, head injury or psychiatric disorder;
* Pregnant women;
* Impaired liver function, abnormal blood coagulation, AIDS, HIV, combine other tumor or special condition;
* Progressive apoplexy;
* With malignant tumors;
* Patients who had participated in other clinical trials within three months prior to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Severity of adverse events | 12 months
  According to National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE)

SECONDARY OUTCOMES:
RA Serology | 1, 3 ,6 and 12 months
  Rheumatoid Factor, C-reactive protein
Disease Activity Score (DAS 28) Index | 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Z Ye, Professor, Principal Investigator — Futian People's Hospital
Locations (1):
- The Fourth People's Hospital of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided